CLINICAL TRIAL: NCT01785719
Title: Ultrasound Characterization of Ovarian Follicle Dynamics During Weight Loss
Brief Title: Evaluation of Ovarian Morphology and Function in Overweight Women During Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Nutrisystem, Inc. (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OSP 69298; R56HD089962 (NIH); R01HD093748-01 (NIH)
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Weight Loss; Anovulation; Amenorrhea; Infertility
Keywords: Weight Loss; Polycystic Ovary Syndrome (PCOS); Ovarian Follicle Development; Metabolism
MeSH Terms: conditions — Weight Loss; Anovulation; Amenorrhea; Infertility; Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: The researchers plan to recruit two cohorts of obese women to the study: (1) those with irregular menstrual cycles and/or PCOS and (2) those with regular menstrual cycles. Both of the cohorts will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overweight Women (Experimental): Regardless of reproductive history, each participant will be provided with six months of the commercial weight loss program, Nutrisystem® D. Nutrisystem® D is a portion-controlled, low calorie, and low glycemic index meal delivery system that provides 1250-1500 kcal/day. It has been proven to help overweight adults achieve real and sustainable weight loss results. When meals and snacks are consumed as instructed, average weight loss is 1-2 lbs per week or 15-20% body weight by the end of six months. Nutrisystem® D offers a balanced meal plan that is consistent with the nutrition recommendations of the USDA for Americans and American Diabetes Association. Each participant will be encouraged to take a daily multivitamin to help meet her micronutrient needs on the program.
  Interventions: Behavioral: Commercial Weight Loss Program

INTERVENTIONS:
Behavioral: Commercial Weight Loss Program — Regardless of reproductive history, each participant will be provided with six months of the commercial weight loss program, Nutrisystem® D. Nutrisystem® D is a portion-controlled, low calorie, and low glycemic index meal delivery system that provides 1250-1500 kcal/day. It has been proven to help overweight adults achieve real and sustainable weight loss results. When meals and snacks are consumed as instructed, average weight loss is 1-2 lbs per week or 15-20% body weight by the end of six months. Nutrisystem® D offers a balanced meal plan that is consistent with the nutrition recommendations of the USDA Dietary Guidelines for Americans and American Diabetes Association. Each participant will be encouraged to take a daily multivitamin to help meet her micronutrient needs on the program.

SUMMARY:
The objective of this study is to explore the effects of weight loss on body composition, metabolic status, reproductive hormones, and ovarian follicle development in obese women with regular menstrual cycles versus obese women with irregular menstrual cycles and/or polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a complex endocrine condition that impacts one in ten women of reproductive age worldwide. It is characterized by a collection of signs and symptoms, including: (1) oligo- or anovulation, (2) hyperandrogenism, and (3) polycystic ovarian morphology. Because obesity worsens the reproductive and metabolic features of the condition, lifestyle intervention aimed at weight loss is recommended as the first-line therapy in overweight / obese patients. Many studies have shown that modest weight loss (5-10%) can improve symptomology in women with PCOS. Yet, the mechanism whereby weight loss might stimulate ovulation or restore menstrual cyclicity remains unclear.

Hence, the goal of this study is to explore the effects of weight loss on body composition, metabolic status, reproductive hormones, and ovarian follicle development in obese women with regular menstrual cycles versus obese women with irregular menstrual cycles and/or PCOS. The researchers believe that a hypocaloric and low-glycemic index eating pattern, based on the nutrition recommendations of the USDA Dietary Guidelines for Americans and American Diabetes Association, will reduce endocrine and metabolic disturbances and consequently improve ovulatory and menstrual cyclicity in PCOS.

To accomplish this objective, the researchers plan to recruit up to 50 obese (i.e. body mass index >30 kg/m*m) women with regular menstrual cycles and up to 50 obese women with irregular menstrual cycles and/or PCOS. Exclusion criteria will include ages <18 or >35 y and the use of hormonal contraception, fertility therapy, or insulin-sensitizing medication in the three months prior to enrollment. This study entails one month of data collection during a baseline interval (Month 1) and six months of data collection during a commercial weight loss program (Nutrisystem® D; Month 2 thru Month 7).

Participants will be evaluated every other day (in Months 1 and 7) or twice per week (in Months 2 thru 6) by transvaginal ultrasonography and venipuncture. Ultrasound images of the ovaries will be assessed for the total number and diameter of individual follicles. Serum samples will be assessed for follicle-stimulating hormone, luteinizing hormone, estradiol, and progesterone. Participants will also be evaluated at up to four time points using multiple metabolic and behavioral tests. Time points of interest will include: (1) Month 1 (i.e. pre-intervention), (2) after 5% weight loss, (3) after 10% weight loss, and (4) Month 7 (i.e. post-intervention). Assessments and endpoints of interest will include: (1) fasting blood tests (to detect serum androgens and markers of metabolic syndrome); (2) an oral glucose tolerance test (to characterize glucose and insulin dynamics at 0, 30, 60, 90, and 120-minutes post-glucose ingestion); (3) a physical examination (to measure height, weight, waist and hips circumference, blood pressure, heart rate, and hirsutism score); (4) a dual x-ray absorptiometry scan (to quantify total and regional fat and lean mass); and (5) a quality of life questionnaire (to evaluate health-related quality of life).

To evaluate further changes in ovarian morphology, reproductive hormones, metabolic status, and body composition after the intervention, participants will be invited to return to the research unit six months after the study ends. The aforementioned procedures (transvaginal ultrasound scan; fasting blood tests; oral glucose tolerance test; physical examination; dual x-ray absorptiometry scan; and quality of life questionnaire) will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.0 kg/m*m.
* Self-reported history of regular menstrual cycles, irregular menstrual cycles, or PCOS.
* Absence of hormonal contraception, fertility therapy, or insulin-sensitizing medication in the three months prior to enrollment.

Exclusion Criteria:

* Pregnant, breastfeeding, or lactating
* Lack of one or both ovaries and/or uterus
* Previous diagnosis of bleeding disorder(s) or current use of blood thinners/anticoagulants
* Vegan or gluten free
* Soy or peanut allergy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-01; Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla Lujan, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University - Human Metabolic Research Unit, Ithaca, New York, United States

REFERENCES:
- [Derived] Carter FE, Jarrett BY, Lee ND, Zaman N, Reich AM, Wilson KA, Oldfield AL, Vanden Brink H, Lujan ME. Changes in antral follicle dynamics following weight loss in women with polycystic ovary syndrome. Hum Reprod. 2025 Nov 1;40(11):2161-2171. doi: 10.1093/humrep/deaf169. PMID 40929646
- [Derived] Oldfield AL, Carter FE, Reeves RE, Jarrett BY, Vanden Brink H, Lujan ME. Impact of a hypocaloric dietary intervention on antral follicle dynamics in eumenorrheic women with obesity. Hum Reprod. 2024 Apr 3;39(4):801-811. doi: 10.1093/humrep/deae017. PMID 38335228
- [Derived] Oldfield AL, Vanden Brink H, Carter FE, Jarrett BY, Lujan ME. Obesity is associated with alterations in antral follicle dynamics in eumenorrheic women. Hum Reprod. 2023 Mar 1;38(3):459-470. doi: 10.1093/humrep/dead007. PMID 36708012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women ages 18-38 with BMI >25 kg/m*m with regular menstrual cycles or irregular menstrual cycles (with or without PCOS). No use of hormonal contraception, fertility therapy, or insulin-sensitizing medication in the 3 months prior to enrollment. All participants completed 4-week baseline evaluation. Participants enrolled before 2018 completed a 12-week hypocaloric dietary intervention. The study was amended in 2018 to increase the duration of the intervention to 24 weeks.
Pre-assignment Details: Most participants experienced a lag between enrollment and the start of baseline due to scheduling, med washout, and/or stage of menstrual cycle. Some participants were lost to follow-up during this time. Additionally, the first 2 weeks of baseline were used to assess ovarian ultrasound image quality and vein status to confirm eligibility. Participants were excluded if we could not achieve consistent high quality ovarian ultrasound images and/or successful venipuncture in the first 2 weeks.
Groups:
- Irregular Cycles (With or Without Additional Features of PCOS): Individuals with irregular menstrual cycles at baseline with or without additional features of PCOS. Irregular menstrual cycles were defined as mean cycle length >35 days over the past year, based on self-reported menstrual cycle dates at enrollment.
- Regular Cycles: Individuals with regular menstrual cycles at baseline. Regular menstrual cycles were defined as mean cycle length 21-35 days over the past year, based on self-reported menstrual cycle dates at enrollment.
Period: 4-week Baseline Evaluation
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Started | 42 | 37
Completed | 34 | 24
Not Completed | 8 | 13
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Poor vein access and/or ultrasound image quality | 4 | 8
Not completed — Exclusionary medication | 2 | 0
Period: Hypocaloric Dietary Intervention
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Started | 34 | 24
Completed | 30 | 18
Not Completed | 4 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Investigator - Poor Compliance | 1 | 2
Not completed — Research Restrictions (COVID) | 1 | 2
Not completed — Poor vein access and/or ultrasound image quality | 0 | 1
Not completed — Participant initiated an exclusionary medication. | 0 | 1
Period: 6-month Post-intervention Follow-up
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Started | 30 | 18
Completed | 18 | 14
Not Completed | 12 | 4
Not completed — Lost to Follow-up | 12 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Exclusionary medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: This table includes baseline characteristics for all participants who completed either the 12-wk or 24-wk hypocaloric dietary intervention, depending on date of enrollment (the study was amended in 2018 to increase the duration of the dietary intervention from 12 to 24 weeks). Regular menstrual cycles were defined as 21-35 days based on self-reported menstrual cycle data from the year leading up to enrollment.
Groups:
- Irregular Cycles (With or Without Additional Features of PCOS): Participants who completed the hypocaloric dietary intervention* and reported irregular menstrual cycles at baseline. Irregular menstrual cycles were defined as mean cycle length >35 days over the past year, based on self-reported menstrual cycle dates at enrollment.
  *Participants enrolled before 2018 completed a 12-week dietary intervention and participants enrolled 2018 and later completed a 24-week dietary intervention.
- Regular Cycles: Participants who completed the hypocaloric dietary intervention* and reported regular menstrual cycles at baseline. Regular menstrual cycles were defined as mean cycle length 21-35 days over the past year, based on self-reported menstrual cycle dates at enrollment.
  *Participants enrolled before 2018 completed a 12-week dietary intervention and participants enrolled 2018 and later completed a 24-week dietary intervention.
- Total: Total of all reporting groups
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles | Total
Number analyzed (Participants) | 30 | 18 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5) | 31 (3) | 29 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 18 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 24 | 17 | 41
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 16 | 39
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 18 | 48
Body Mass Index [Mean (Standard Deviation); unit: kg/m*m] | 37 (6) | 37 (7) | 37 (6)
Menstrual Cycle Length [Mean (Standard Deviation); unit: days] | 84 (67) | 30 (2) | 65 (59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Ovulatory/Menstrual Function
Description: Participants with irregular menstrual cycles at baseline were categorized as "responders" or "non-responders" based on any changes they experienced in menstrual cyclicity over the course of the intervention. "Responders" were defined as participants who shifted towards a more favorable menstrual cycle status over the course of the intervention. "Non-responders" were defined as participants who experienced no change or a shift to a less favorable menstrual cycle status over the course of the intervention. Menstrual cycle status categories were defined as "Amenorrhea" (mean cycle length>90 days; least favorable), "Oligomenorrhea" (mean cycle length 36-90 days; unfavorable), and "Regular" (mean cycle length 21-35 days; most favorable). All participants with regular menstrual cycles at baseline maintained regular cycles over the course of the intervention and were therefore not included in this analysis.
Time Frame: Up to 7 months
Population: This table includes outcome data for all participants who completed either the 12-wk or 24-wk hypocaloric dietary intervention, depending on year of enrollment (participants pre-2018 completed 12 weeks, participants 2018 and later completed 24 weeks). Irregular menstrual cycles were defined as mean cycle length >35 days over the past year, based on self-reported menstrual cycle dates at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS)
Number analyzed (Participants) | 30
Participants
  Responders | 12
  Non-Responders | 18

2. Secondary Outcome: Change From Baseline Follicle Number Per Ovary
Description: Change in follicle number per ovary (FNPO) from baseline to the end of a hypocaloric dietary intervention. Ovarian images were collected using 3D transvaginal ultrasonography and were assessed for morphological endpoints by trained raters using the 2D offline grid method. FNPO was calculated by summing all 2-9 mm follicles in each ovary. Left and right FNPO were averaged for each participant before baseline to post-intervention changes were calculated.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Follicle number per ovary
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
Follicle number per ovary | -5 (14) | -9 (11)

3. Secondary Outcome: Change From Baseline Reproductive Hormones
Description: Change in reproductive hormones from baseline to the end of a hypocaloric dietary intervention. Blood samples were collected in the morning after an overnight fast during the early follicular phase as confirmed by the absence of a dominant follicle or corpus luteum on ultrasound. Hormones reported include:
  * Total testosterone: Evaluated by the Brigham Research Assay Core (Harvard) using liquid chromatography tandem mass-spectrometry. Results are reported in ng/dL.
  * Anti-Müllerian hormone (AMH): Evaluated using the Motive Biosciences (formerly Ansh Labs) picoAMH ELISA. Results are reported in ng/mL
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
ng/dL
  Change in Total testosterone (ng/dL) | 20 (52) | -5 (8)
  Change in AMH (ng/dL) | 0.32 (2.77) | -0.38 (2.91)

4. Secondary Outcome: Change From Baseline Metabolic Status (HOMA-IR)
Description: Change in metabolic status from baseline to the end of a hypocaloric dietary intervention. HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) was used as an indicator of metabolic status. HOMA-IR uses fasting blood glucose and insulin values to approximate insulin resistance. Blood glucose and insulin were measured in the morning after an overnight fast during the early follicular phase as confirmed by the absence of a dominant follicle or corpus luteum on ultrasound. HOMA-IR was calculated by multiplying blood glucose (mg/dL) by insulin (mIU/mL) and dividing by 405. A higher HOMA-IR score is indicative of increased insulin resistance.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
HOMA-IR score | -1.3 (2.5) | -0.9 (0.8)

5. Secondary Outcome: Change From Baseline Total Percent Body Fat
Description: Change in total percent body fat from baseline to the end of a hypocaloric dietary intervention. Body fat was measured using the Hologic Discovery A Dual X-Ray Absorptiometry (DXA) Scanner.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent body fat
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
Percent body fat | -1.8 (1.6) | -1.6 (4.3)

6. Secondary Outcome: Change From Baseline Ovarian Volume
Description: Change ovarian volume (cm^3) from baseline to the end of a hypocaloric dietary intervention. Ovarian images were collected using 3D transvaginal ultrasonography and were assessed for morphological endpoints by trained raters using the 2D offline grid method. Ovarian volume was calculated using a modified formula for a prolate ellipsoid. Left and right ovarian volumes were averaged for each participant before baseline to post-intervention changes were calculated.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
cm^3 | -1.9 (2.8) | 0.9 (2.0)

7. Secondary Outcome: Change From Baseline Free Androgen Index (FAI)
Description: Change in FAI from baseline to the end of a hypocaloric dietary intervention. Blood samples were collected in the morning after an overnight fast during the early follicular phase as confirmed by the absence of a dominant follicle or corpus luteum on ultrasound. Free Androgen Index (FAI) is the ratio of total testosterone to sex hormone binding globulin (SHBG), indicating the amount of active testosterone in the blood. SHBG was evaluated by the Cornell Human Nutrition Chemistry Service Laboratory using Immulite 2000 immunoassay. FAI levels of 5 or higher are indicative of PCOS.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: free androgen index
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
free androgen index | 2 (9) | -1 (1)

8. Secondary Outcome: Change From Baseline BMI
Description: Change in BMI from baseline to the end of a hypocaloric dietary intervention.
Time Frame: Up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
Number analyzed (Participants) | 30 | 18
kg/m^2 | -2.8 (1.5) | -3.8 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 13 months (including up to 7 months of baseline and dietary intervention, plus a single follow-up visit 6 months later).
Description: All participants who enrolled in the study were considered at risk for adverse events. A systematic approach was used to assess adverse events. During each study visit (2-6 times per week), research team members asked participants whether they were experiencing any adverse symptoms related to the study diet or study procedures. Research team members reviewed fasting blood glucose results and did not proceed with the oral glucose tolerance test if a participant's value exceeded 120 mg/dL.
Arm/Group | Irregular Cycles (With or Without Additional Features of PCOS) | Regular Cycles
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/37
Other Adverse Events (participants affected / at risk) | 10/42 | 2/37
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Irregular Cycles (With or Without Additional Features of PCOS) (N=42) | Regular Cycles (N=37)
Fasting blood glucose value of >120 mg/dL (Endocrine disorders) | 3 (3) | 0 (0) — Participant exhibited an elevated fasting blood glucose (>120 mg/dL), which disqualified them from participating in the oral glucose tolerance test. The participant was advised to share the fasting blood glucose results with their medical provider.
2 hour blood glucose value of 140-199 mg/dL (Endocrine disorders) | 6 (8) | 1 (1) — Participant had normal fasting blood glucose and proceeded with 2-hr 75g glucose tolerance test. The participant's 2-hour blood glucose was between 140-199 mg/dL, consistent with impaired glucose tolerance. Participant was advised to alert provider.
Hypertrophic scarring at venipuncture site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant experienced hypertrophic scarring at the venipuncture site after 1 month of study participation.
Bloating and gastrointestinal discomfort (Metabolism and nutrition disorders) | 1/34 (1) | 0/24 (0) — Participant experienced bloating and gastrointestinal discomfort during their first two weeks consuming the study diet (Nutrisystem D).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT01785719/Prot_ICF_006.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT01785719/SAP_004.pdf